CLINICAL TRIAL: NCT06348576
Title: A Multicenter, Randomized, Double-blind, Active-control, Phase III Study to Evaluate the Efficacy and Safety of AD-209 in Patients With Essential Hypertension
Brief Title: Phase III Study to Evaluate the Efficacy and Safety of AD-209
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Addpharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AD-209P3
Record Dates: First submitted 2024-04-01; First posted 2024-04-04 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Hypertension,Essential
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): AD-209+AD-2091 Placebo
  Interventions: Drug: AD-209; Drug: AD-2091 Placebo
- Control group (Active Comparator): AD-2091+AD-209 Placebo
  Interventions: Drug: AD-2091; Drug: AD-209 Placebo

INTERVENTIONS:
Drug: AD-209 — PO, Once daily(QD), 8weeks
  Arms: Test group
Drug: AD-2091 — PO, Once daily(QD), 8weeks
  Arms: Control group
Drug: AD-209 Placebo — PO, Once daily(QD), 8weeks
  Arms: Control group
Drug: AD-2091 Placebo — PO, Once daily(QD), 8weeks
  Arms: Test group

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of AD-209

DETAILED DESCRIPTION:
Condition or disease : hypertension

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Other inclusions applied

Exclusion Criteria:

* Orthostatic hypotension with symptom
* Other exclusions applied

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Change rate of MSSBP | Baseline, Week 8
  Change from baseline in mean sitting systolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Chang Gyu Park, M.D., Ph.D, Principal Investigator — Korea University Guro Hospital
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No